CLINICAL TRIAL: NCT03693196
Title: The Effect of Different Dental Implant Surface Characteristics on Bone Immunological Biomarkers and Microbiological Parameters: A Randomized Clinical Study
Brief Title: The Effect of Different Dental Implant Surface Characteristics on Immunological and Microbiological Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, BİLGE KARCI, Research assistant, Necmettin Erbakan University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2016/009
Record Dates: First submitted 2018-05-07; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Peri-implant Mucositis; Peri-Implantitis
Keywords: Dental implant; Immunology; Microbiology; Surface characteristic
MeSH Terms: conditions — Peri-Implantitis | interventions — Demography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Straumann® (Other): Titanium implants the surfaces of which were roughened with SLA (sandblasted and acid-etched titanium surface) (Straumann®, Basel, Sweden). Immunological parameters (PICF, Perio-paper®) , microbiological parameters of peri-implantitis (subgingival plaque, Hu-Friedy®), demographic and clinical periodontal measurements (Williams probe, PCPNU-15 Hu-Friedy®) were compared between groups.
  Interventions: Other: PICF, Perio-paper®; Other: Subgingival Plaque, Hu-Friedy®; Other: Williams probe, PCPNU-15 Hu-Friedy®; Other: Demographic
- Astra Tech, OsseoSpeed™ (Other): Implants the surfaces of which were roughened by modifying with fluorine (Astra Tech, OsseoSpeed™, Sweden). Immunological parameters (PICF, Perio-paper®), microbiological parameters of peri-implantitis (subgingival plaque, Hu-Friedy®), demographic and clinical periodontal measurements (Williams probe, PCPNU-15 Hu-Friedy®) were compared between groups.
  Interventions: Other: PICF, Perio-paper®; Other: Subgingival Plaque, Hu-Friedy®; Other: Williams probe, PCPNU-15 Hu-Friedy®; Other: Demographic
- Nobel Biocare, Replace® (Other): Implants the surfaces of which were roughened by anodization (TiUnite Nobel Biocare, Replace® Conical Connection, Sweden). Immunological parameters (PICF, Perio-paper®), microbiological parameters of peri-implantitis(subgingival plaque, Hu-Friedy®), demographic and clinical periodontal measurements (Williams probe, PCPNU-15 Hu-Friedy®) were compared between groups.
  Interventions: Other: PICF, Perio-paper®; Other: Subgingival Plaque, Hu-Friedy®; Other: Williams probe, PCPNU-15 Hu-Friedy®; Other: Demographic

INTERVENTIONS:
Other: PICF, Perio-paper® — PICF was collected from the mesio-buccal area of the implant by using paper tapes. Paper tapes were placed 1-2 mm inside the peri-implant sulcus by using a dental tweezer. After they were kept for 30 s, the paper tapes were placed in sterile microcentrifuge tubes which contained 200 µL phosphate-buffered saline (PBS). The tubes were kept at -80°C until the analysis day. TNF-α, PGE2, RANKL, RANK, and OPG, which are immunological markers of peri-implant disease were compared between groups.
Other: Subgingival Plaque, Hu-Friedy® — Subgingival plaque samples were collected about 15 min after PICF was collected. Supragingival plaque was carefully removed by using a sterile scale. Implants were isolated using cotton rolls and dried with an air spray. Subgingival plaque samples were collected from the mesio-buccal area of the implant by using sterile plastic Gracey curettes during 30 s (Hu-Friedy). The samples collected were transferred to sterile microcentrifuge tubes containing 200 µL PBS. The tubes were kept at -80°C until the analysis day. Porphyromonas gingivalis, Treponema denticola, Tannerella forsythia, Fusobacterium nucleatum, Prevotella intermedia, and Streptococcus oralis, which are microbiological agents of peri-implantitis were compared between groups.
Other: Williams probe, PCPNU-15 Hu-Friedy® — Clinical periodontal measurements were recorded using Williams probe. The plaque index, gingival index, pocket depth, bleeding on probing, clinical attachment level, and keratinised tissue width around the implant were recorded. The implants included were categorised into three groups, namely, healthy, peri-implant mucositis, and peri-implantitis. Panoramic radiographs were acquired to assess the interproximal bone levels around the implant.
Other: Demographic — Age, gender and state of smoking were compared between groups.

SUMMARY:
Objectives: To assess the levels of TNF-α, PGE2, RANKL, RANK, OPG, which are immunological markers of peri-implant disease and F. nucleatum, P. gingivalis, T. denticola, T. forsythia, P. intermedia, S. oralis, which are microbiological agents of peri-implantitis, in areas where SLA, fluorine-modified and anodized implant surfaces are used.

Material and methods: In this study, 71 implants of 37 patients were assessed. The patients were grouped according to the surface characteristics of the implants. Group 1: SLA surface, Group 2: Fluorine modifying surface, Group 3:Anodization surface Plaque index (PI), gingival index (GI), bleeding on probing (BOP), pocket depths (PD), clinical attachment levels (CAL) and keratinized tissue width (KTW) were measured. Peri-implant sulcus fluid and subgingival plaque samples were collected.

Results: PI was found to be significantly lowest in Group 1, higher in Group 3. Group 3 implants were found to have more bleeding on probing significantly. It was found to be higher peri-implant mucositis and peri-implantitis in Group 3. GI, PD, CAL, KTW were not found to differ between groups. No significant differences were found between TNF-α, PGE2, RANKL, RANK, OPG. While F. nucleatum, T. forsythia, T. denticola and P. intermedia were found to be significant highest in Group 3, P. gingivalis and S. oralis were found to be high in Group 2.

Conclusion: Peri-implantitis rate, BOP and PI were found to be higher in Group 3. F. nucleatum, T. forsythia, T. denticola, and P. intermedia were found to be significantly high in Group 3 implants. This situation can be associated with the porous structure of anodized surface.

DETAILED DESCRIPTION:
1. | INTRODUCTION Dental implants are commonly used in partly and completely edentulous patients in order to improve function, aesthetic appearance and life quality. Successful osseointegration is provided with recently developed surface modifications. Some of these are SLA (Sand-blasted, Largegrit, Acid-etched), fluorine modified surface and anodized surfaces. SLA implants are obtained by spraying large sand grits on the implant. Modification of dental implants with fluorine is a chemical method in which fluorine, one of the basic elements of bone, is added on the surface to increase osteogenesis. Implants with anodized surface form with micro or nano porous surfaces as a result of high intensity (200 A/m2) or potential (100 V) potansiostatic or galvanostatic anodization of titanium inside strong acids such as H2SO4, H3PO4, HNO3, HF. When this application is compared with passivated surfaces, it results in the thickening of titanium oxide layer.

   The objective of this study is to assess comparatively the levels of TNF-α, PGE2, RANKL, RANK, OPG, which are immunological markers of peri-implant disease and Porphyromonas gingivalis (P. gingivalis), Treponema denticola (T. denticola), Tannerella forsythia (T. forsythia), Fusobacterium nucleatum (F. nucleatum), Prevotella intermedia (P. intermedia), Streptococcus oralis (S. oralis), which are microbiological agents of peri implantitis, in areas where SLA, fluorine-modified and anodized implant surfaces are used.
2. | MATERIAL AND METHODS 2.1 | Study Population The study was conducted by calling back patients whose partial missing teeth were treated with implant supported fixed restorations at Necmettin Erbakan University Faculty of Dentistry, Department of Periodontology and whose implants had been functioning for at least a year. The inclusion criteria of the study were not having any systemic disorders that can affect bone metabolism and wound healing, being older than 18, having prostheses in the posterior area, having received cement retained implant prosthesis in which standard abutment was used, having implant prosthesis which had been functioning for at least a year, not having received bone augmentation procedure or advanced implant surgery during implant surgery, not having received periodontal treatment during the previous year, and having received one of SLA, fluorine modified or anodized implants. The exclusion criteria were uncontrolled diabetes mellitus and other uncontrolled diseases, pregnancy, lactation, aggressive periodontitis, overdenture patients and parafunctional habits such as bruxism. In the study, 71 implants of 37 patients, 24 females and 13 males, were assessed. The patients called were grouped in three according to the surface characteristics of the implants.

Group 1: Titanium implants the surfaces of which were roughened with SLA (sandblasted and acid-etched titanium surface) (Straumann®, Basel, Sweden), Group 2: Implants the surfaces of which were roughened by modifying with fluorine (Astra Tech, OsseoSpeed™, Sweden) Group 3: Implants the surfaces of which were roughened by anodization (TiUnite Nobel Biocare, Replace® Conical Connection, Sweden).

The implants included were grouped in three as healthy, peri-implant mucositis and peri-implantitis. Peri-implantitis group included implants which had bleeding and/or supuration at probing, pocket depth > 4 mm at least in one area and 2 mm or more radiographic bone loss around the implant, peri-implant mucositis group included implants which had bleeding and/or supuration at probing and no radiographic bone loss around the implant and the healthy group included implants which did not have inflammation around the implant, bleeding or supuration at probing and radiograph bone loss around the implant.

2.2 | Clinical Periodontal Measurements The indexes and measurements used in the study were measured within a specific order and recorded in data recording forms prepared according to this order. Plaque index (PI), gingival index (GI), pocket depths (PD), bleeding on probing, clinical attachment levels (CAL) and keratinized tissue width around the implant (KTW) were recorded. Panoramic radiographs were taken to assess the interproximal bone levels around the implant (Morita, Veraviewepocs 3D F40, Japan).

2.3 | Collecting the Peri-implant crevicular fluid (PICF) and Subgingival Plaque Samples After taking PI from all individuals, plaques and soft additions around the implant were removed and after the area was isolated with the help of cotton rolls, the teeth were dried with air. PICF was collected from the mesio-buccal area of the implant by using paper tapes (Perio-paper, Oraflow Inc, New York, USA). Subgingival plaque samples were collected about 15 minutes after PICF was collected.

2.4 | PICF analysis Commercial enzyme-linked immunosorbent assay (ELISA) kits were purchased for the measurement of TNF-α, PGE2, RANKL, RANK, OPG and assays were carried out according to the manufacturers' recommendations (Elabscience Biotechnology Co.,Ltd, Wuhan, China).

2.5 | Preparation and Assessment of Genomic DNA Forthe DNA extraction, the collected subgingival plaque samples were processed using a commercially available kit (GF-1 bacterial DNA extraction kit, Vivantis, Malaysia) according to the instructions of the manufacturer.

2.6 | Real-Time Quantitative Polymerase Chain Reaction Selected putative periodontal pathogens (P. intermedia, T. forsythia, T.denticola, F. nucleatum, P.gingivalis, Streptococcus oralis) and total bacterial load in the subgingival biofilms were detected as described previously.

2.7 | Statistical Analysis SPSS 19.0 (IBM Inc., Chicago, IL, USA) program was used for the statistical analyses of the study. Normality test for continuous numerical variables was conducted with Kolmogorov-Smirnov analysis method. Since all of the variables were not normally distributed, non-parametrical methods were preferred in the analyses. Mann-Whitney U method was preferred for two independent groups, while Kruskal-Wallis was used for multiple groups. p<0,05 was accepted statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* not having any systemic disorders that can affect bone metabolism and wound healing,
* being older than 18,
* having prostheses in the posterior area,
* having received cement retained implant prosthesis in which standard abutment was used,
* having implant prosthesis which had been functioning for at least a year,
* not having received bone augmentation procedure or advanced implant surgery during implant surgery,
* not having received periodontal treatment during the previous year,
* having received one of SLA, fluorine modified or anodized implants.

Exclusion Criteria:

* uncontrolled diabetes mellitus and other uncontrolled diseases,
* pregnancy,
* lactation,
* aggressive periodontitis,
* overdenture patients
* parafunctional habits such as bruxism.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Real-time polymerase chain reaction (PCR) | an average of 1 year
  For DNA extraction, the collected subgingival plaque samples were processed using a commercially available kit (GF-1 bacterial DNA extraction kit, Vivantis, Malaysia) according to the manufacturer's instructions. Selected putative periodontal pathogens and total bacterial load in the subgingival biofilms were detected as described previously.

SECONDARY OUTCOMES:
Commercial enzyme-linked immunosorbent assay (ELISA) kits | an average of 1 year
  ELISA kits were purchased for measuring TNF-α, PGE2, RANKL, RANK, and OPG, and assays were carried out according to the manufacturers' recommendations (Elabscience Biotechnology Co., Ltd, Wuhan, China).

CONTACTS AND LOCATIONS:
Overall Officials: Elif Öncü, Study Director — Necmettin Erbakan University, Faculty of Dentistry, Department of Periodontology, Konya, Turkey; Metin Doğan, Study Chair — Necmettin Erbakan University, Meram Faculty of Medicine, Department of Microbiology, Konya, Turkey

REFERENCES:
- [Background] Gurlek O, Gumus P, Nile CJ, Lappin DF, Buduneli N. Biomarkers and Bacteria Around Implants and Natural Teeth in the Same Individuals. J Periodontol. 2017 Aug;88(8):752-761. doi: 10.1902/jop.2017.160751. Epub 2017 Apr 25. PMID 28440740
- [Background] Le Guehennec L, Soueidan A, Layrolle P, Amouriq Y. Surface treatments of titanium dental implants for rapid osseointegration. Dent Mater. 2007 Jul;23(7):844-54. doi: 10.1016/j.dental.2006.06.025. Epub 2006 Aug 14. PMID 16904738
- [Background] Mombelli A, Decaillet F. The characteristics of biofilms in peri-implant disease. J Clin Periodontol. 2011 Mar;38 Suppl 11:203-13. doi: 10.1111/j.1600-051X.2010.01666.x. PMID 21323716
- [Result] Derks J, Hakansson J, Wennstrom JL, Tomasi C, Larsson M, Berglundh T. Effectiveness of implant therapy analyzed in a Swedish population: early and late implant loss. J Dent Res. 2015 Mar;94(3 Suppl):44S-51S. doi: 10.1177/0022034514563077. Epub 2014 Dec 11. PMID 25503901
- [Result] Derks J, Schaller D, Hakansson J, Wennstrom JL, Tomasi C, Berglundh T. Effectiveness of Implant Therapy Analyzed in a Swedish Population: Prevalence of Peri-implantitis. J Dent Res. 2016 Jan;95(1):43-9. doi: 10.1177/0022034515608832. PMID 26701919
- [Result] Shibli JA, Melo L, Ferrari DS, Figueiredo LC, Faveri M, Feres M. Composition of supra- and subgingival biofilm of subjects with healthy and diseased implants. Clin Oral Implants Res. 2008 Oct;19(10):975-82. doi: 10.1111/j.1600-0501.2008.01566.x. PMID 18828812